CLINICAL TRIAL: NCT04755361
Title: Examining the Effectiveness of a Critical Time Intervention to Stabilize Trajectories Out of Homelessness for Youth
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: LOFT Community Services (Other); Covenant House Toronto (Other); Wellesley Institute (Unknown)
Responsible Party: Principal Investigator, Sean Kidd, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 162/2020
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Homeless Persons

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Housing Outreach Project - Collaboration (HOP-C) + Treatment as Usual (Experimental): The treatment condition is HOP-C plus treatment as usual (TAU).
  Interventions: Behavioral: Housing Outreach Project Collaboration (HOP-C)
- Treatment As Usual (No Intervention): TAU for this population reflects the standard array of services accessed by transitional youth populations. Most will have some contact with a youth worker with ranging focus and intensity (none likely to receive case management at HOP-C intensity), and very few will have any routine contact with other professionals or peer support. They may have some sporadic access to skills development programs and primary healthcare providers with mental health and addictions needs addressed primarily through emergency services at times of crisis.

INTERVENTIONS:
Behavioral: Housing Outreach Project Collaboration (HOP-C) — HOP-C has several components: HOP-C Case management is outreach-based (emphasizing community and home contacts) and participant goal-driven, providing coaching and skill building in key functional domains and assistance with navigating various systems (justice, housing, employment, health, education). The mental health component has two parts. One is a weekly, 90-minute, mental health and wellness-oriented group. The group acts, for most, as a stepped care approach, with members moving on to access individual psychotherapy as needed. Peer support is provided by youth with a history of lived experience of homelessness who have successfully achieved housing stability and progress in major life domains. Peers receive extensive training and are formally hired into these roles with their being 2-3 peers on the team.
  Arms: Housing Outreach Project - Collaboration (HOP-C) + Treatment as Usual

SUMMARY:
Problem Statement: This proposal addresses the problem of youth not being adequately supported as they attempt to transition out of homelessness. This problem leads to frequent cycling in and out of homelessness, protracted periods of homelessness, and increased exposure to an array of serious risks to health and wellbeing. This is not just an issue of housing. While adequate housing is necessary to youth exiting homelessness it is not, in and of itself, sufficient to ensure success in sustaining housing nor flourishing as a result of housing.

Objective: This proposal tests a complex, critical time intervention for youth in transition out of homelessness. This intervention, which is team-based and comprised of integrated case management, peer support, and mental health supports, has proven feasible in pilot and feasibility trials. Its objective is to stabilize housing trajectories and improve outcomes in major life domains.

Specific Aims: The primary aim of this study is to determine if the provision of 1 year of the critical time intervention HOP-C can improve the outcomes of youth who have transitioned into stable housing in the past 6 months. It is hypothesized that, compared with treatment as usual, housing, employment, education, and mental health outcomes will be significantly better for youth who receive HOP-C and that these gains will be sustained. Changes in quality of life, social supports, and psychological wellbeing will be explored as secondary outcomes.

Partners: This study builds on a partnership between the Centre for Addiction and Mental Health (research capability, mental health service expertise) and two established Toronto service providers focusing on homeless youth populations (Covenant House - Toronto; LOFT Community Services).

Study Design: This study is a single blind, randomized controlled trial comparing the outcomes of the transitional intervention described above with typical supports provided in the community. Assessments will be conducted at baseline, mid-point (6 months), post-intervention (1 year), and at 6 months follow up.

Implications: From a trial design perspective, the proposed study would provide evidence supporting a rationale for future trials and wide implementation. Pending positive outcomes, this would flow into multisite trial and implementation grant applications and further collaborations with others working within Canada and elsewhere. More broadly, this line of investigation has synergy with the increasingly larger and better-organized movements towards addressing homelessness in Canada. These efforts have included At Home/Chez soi - the largest study to date of housing first and Making the Shift, an NCE-funded collaborative effort towards ending youth homelessness in Canada. Collectively, these developments (in which the applicants are substantively involved), present the opportunity for both scaling the critical time intervention proposed here and its ultimately being combined with other approaches (e.g., housing first, family reunification, support in transitions from protection and justice systems). Such systems-oriented strategies, girded by evidence, hold the greatest promise for ameliorating the problem of youth homelessness and homelessness overall in Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be aged 16-25 (service mandate of participating organizations and captures the age span of youth transitioning from homelessness - in previous studies mean age ranged from 21-22).
2. All participants will have experienced at least 6 months of homelessness defined as being a lack of fixed, regular, and adequate housing across their lifetime.
3. Participants will have been in stable housing for between 1 day and 6 months. This period has characterized the transitional experience in previous research14. Stable housing is a housing arrangement that either (i) involves an individual holding a lease, (ii) is a supported housing arrangement with a tenure of 12+ months, or (iii) involves the person residing with a family member wherein the individual and service provider attest to stability. These broad criteria are necessary due to the diversity of housing arrangements into which youth transition.
4. Proficiency in English.

Exclusion Criteria:

1) Has transitioned to a residence outside of Toronto or plans to do so within the coming year.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Housing Stability | Every 6 months after baseline up to 18 months.
  Housing stability will be assessed using the Residential Time Line Follow-back (RTLFB) inventory. This tool will be used to calculate the percentage of days spent stably housed during each 6-month assessment period - the number of days housed divided by the total number of days. Higher percentages indicate better outcomes.
Education and Vocational Engagement | Every 6 months after baseline up to 18 months.
  Education and vocational engagement will be pooled and assessed using the Residential Time Line Follow-back (RTLFB) inventory. This tool will be used to calculate the percentage of days spent engaged in education or vocational activities during each 6-month assessment period - the number of days engaged divided by the total number of days. Higher percentages indicate better outcomes.

SECONDARY OUTCOMES:
Mental Health Crises | Every 6 months after baseline up to 18 months.
  The secondary outcome is an assessment of mental health crises, operationalized as nights spent in hospital during the assessment time period for any mental health and/or addiction problem. More nights spent indicate worse outcomes.
Self-reported Mental Health | Every 6 months after baseline up to 18 months.
  Self-reported Mental Health will be operationalized as (i) participant ratings on the Colorado Symptom Index which is a 15-item measure of psychiatric symptoms measured on a 5 point scale. Higher scores indicate greater distress.
Quality of Life | Every 6 months after baseline up to 18 months.
  Quality of Life will be measured using the World Health Organization Quality of Life Scale - Bref: WHO QOL Bref, which is a 24 item scale that captures: Physical health with 7 items, psychological health with 6 items, social relationships with 3 items, and environmental health with 8 items. Higher scores indicate better outcomes.
Resilience | Every 6 months after baseline up to 18 months.
  Resilience will be assessed using the Connor-Davidson Resilience Scale. Respondents rate 10 items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4. A higher score indicates higher resilience.
Subjective housing stability | Every 6 months after baseline up to 18 months.
  Subjective housing stability will be assessed with the Housing Security Scale - Version 2 (HSSV2). It is a 21 item scale designed for youth homelessness populations to assess housing stability with higher scores indicating greater stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The plan is to provide de-identified data to other researchers after analyses are complete.
Supporting Information: Study Protocol, SAP
Time Frame: Pending
Access Criteria: Pending

REFERENCES:
- See also: More details on the HOP-C program of work. — https://www.homelesshub.ca/HOP-C